CLINICAL TRIAL: NCT04706637
Title: A Multicenter Randomized Exploratory Clinical Trial to Evaluate the Effect of Bone Metabolism and the Efficacy of Evogliptin and Dapagliflozin for Blood Sugar in the Menopause Female Patients With Osteopenia and Type 2 Diabetes
Brief Title: A Clinical Trial to Evaluate the Bone Metabolism and the Blood Sugar of Evogliptin and Dapagliflozin
Acronym: EVOMETA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVOMETA-04
Record Dates: First submitted 2020-12-29; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Bone Diseases, Metabolic; Diabetes Mellitus, Type 2
Keywords: osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic; Diabetes Mellitus, Type 2 | interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one; dapagliflozin

STUDY DESIGN:
Intervention Model Description: If a subject voluntarily agrees to participate and meets the inclusion and exclusion criteria for the clinical trial, the subject will be randomly assigned to one of the two arms.
  1. Arm 1: evogliptin 5mg + metformin, oral administration once a day for 48 weeks
  2. Arm 2: dapagliflozin 10mg + metformin, oral administration once a day for 48 weeks
Masking Description: The subject will be randomly assigned to one of the two arms. This is an open-label trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- evogliptin (Experimental): evogliptin 5 mg + metformin, oral administration once a day for 48 weeks
  Interventions: Drug: Evogliptin
- dapagliflozin (Active Comparator): dapagliflozin 10mg + metformin, oral administration once a day for 48 weeks
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Evogliptin — evogliptin 5mg + metformin, oral administration once a day for 48 weeks
  Arms: evogliptin
Drug: Dapagliflozin — dapagliflozin 10mg + metformin, oral administration once a day for 48 weeks
  Arms: dapagliflozin

SUMMARY:
This multi-center, randomized and exploratory clinical trial is designed to evaluate the effect of bone metabolism and blood sugar of evogliptin and dapagliflozin in the menopause female patients with osteopenia and type 2 diabetes.

The trial will evaluate bone metabolism (bone markers and bone density) and blood sugar (AGE and glucose variability) after 12 weeks and 48 weeks.

This clinical trial conducts in two arms, and each arm recruits 60 subjects.

DETAILED DESCRIPTION:
This clinical trial is to evaluate the effect of bone metabolism and blood sugar of evogliptin and dapagliflozin in the menopause female patients with osteopenia and type 2 diabetes.

Bone metabolism (bone markers and bone density) and blood sugar (AGE and glucose variability) after 12 weeks and 48 weeks will be evaluated.

This clinical trial conducts in two arms, and each arm recruits 60 subjects. If a subject voluntarily agrees to participate and meets the inclusion and exclusion criteria for the clinical trial, the subject will be randomly assigned to one of the two arms.

The total period after the subject enrollment is 48 weeks, and a total of six visits are made with screening, baseline, 12 weeks, 24 weeks, 36 weeks, and 48 weeks.

Efficacy evaluation will be carried out changes on blood sugar, bone markers and density and after 12 and 48 weeks.

The results of this study are intended to be a reference to future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women between 40 and 70 years of age with type 2 diabetes patients who are not taking diabetes drugs or who are not controlled by blood sugar at 7.0≤HbA1c≤9.0 while taking metformin

   ※ Menopause corresponds when one or more of the following three conditions are satisfied. (1) 12 months of amenorrhea (2) In the case of FSH≥40 mIL(milli-international unit)/mL in women over 50 years who have undergone a hysterectomy or 6 months of amenorrhea (3) Patients 6 weeks after ovariectomy
2. Lumbar, neck of femur and total femur bone density measurements were -2.4≤T-score≤-1.0
3. Obtained written informed consent from a patient
4. Patients who can participate during clinical trials and perform all planned trial procedures and visits.

Exclusion Criteria:

1. A person who has taken a diabetes medications other than metformin within 12 weeks, or who is hypersensitivity to DPP4(dipeptidyl peptidase-4) inhibitors or SGLT2 inhibitors.
2. AST(ASpartate Transaminase) or ALT(ALanine Transaminase) exceeds 2 times the upper limit of the normal range in laboratory tests
3. Patients with moderate or severe renal impairment, end-stage renal disease (ESRD) or dialysis
4. Patients whose eGFR(epidermal growth factor receptor) calculated using MDRD formula within 4 weeks before screening or at screening is less than 60 mL/minute/1.73 m2
5. In the case of osteoporosis medication dosage as follows:

   * Patients who have ever used bisphosphonate formulations
   * Patients who have used female hormones, SERM(Selective Estrogen Receptor Modulator), denosumab, and parathyroid hormone preparations within 12 months
6. Have bone or mineral metabolic diseases or have received treatment that affects them (1) Steroid; - Oral steroid 2.5mg or more has been continuously taken for more than 3 months from the date of consent - Continuous use of systemic or inhaled steroids for more than 3 months from the date of consent (2) Taking diuretics (3) Patients at risk for secondary osteoporosis
7. Patients who have participated in other clinical trials within 3 months
8. Patients with a history of malignant tumors within 5 years
9. Those who have a history of hypersensitivity to the main ingredients and additives of the trial drugs
10. Patients with type 1 diabetes or diabetic ketoacidosis
11. Patients with genetic problems such as galactose intolerance, Lapp deficiency, or glucose-galactose malabsorption
12. Any other patient that the investigator has determined is unsuitable for this clinical trial

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — menopause female patients with osteopenia and type 2 diabetes.
Enrollment: 120 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Change of bone density | Screening, 48 weeks
  Change from screening bone density of lumbar spine 1-4, neck of femur and whole femur at 48 weeks
Change of CTX(C-terminal telopeptide of type I collagen) | Baseline, 12 weeks, 48 weeks
  Change from baseline bone marker CTX(C-terminal telopeptide of type I collagen) at 12 weeks and 48 weeks.
Change of P1NP(Procollagen type 1 Aminoterminal Propeptide) | Baseline, 12 weeks, 48 weeks
  Change from baseline bone marker P1NP(Procollagen type 1 Aminoterminal Propeptide) at 12 weeks and 48 weeks
Change of 25OHD(25 Hydroxyvitamin D) | Baseline, 12 weeks, 48 weeks
  Change from baseline bone metabolism indicator 25OHD(25 Hydroxyvitamin D) at 12 weeks and 48 weeks
Change of PTH(Parathyroid Hormone) Intact | Baseline, 12 weeks, 48 weeks
  Change from baseline bone metabolism indicator PTH(Parathyroid Hormone) Intact at 12 weeks and 48 weeks
Change of FGF23 (Fibroblast growth factor 23) | Baseline, 12 weeks, 48 weeks
  Change from baseline bone metabolism indicator FGF23(Fibroblast growth factor 23) at 12 weeks and 48 weeks
Change of 24 hour urine calcium | Baseline, 12 weeks, 48 weeks
  Change from baseline bone metabolism indicator 24 hour urine calcium at 12 weeks and 48 weeks
Change of 24 hour urine phosphate | Baseline, 12 weeks, 48 weeks
  Change from baseline bone metabolism indicator 24 hour urine phosphate at 12 weeks and 48 weeks
Change of 24 hour urine creatinine | Baseline, 12 weeks, 48 weeks
  Change from baseline bone metabolism indicator 24 hour urine creatinine at 12 weeks and 48 weeks

SECONDARY OUTCOMES:
Change of HbA1C | Baseline, 12 weeks, 48 weeks
  Change from baseline HbA1C at 12 weeks and 48 weeks
Change of FBS(Fasting Blood Sugar) | Baseline, 12 weeks, 48 weeks
  Change from baseline FBS(Fasting Blood Sugar) at 12 weeks and 48 weeks
Change of insulin | Baseline, 12 weeks, 48 weeks
  Change from baseline insulin at 12 weeks and 48 weeks
Change of c-peptide | Baseline, 12 weeks, 48 weeks
  Change from baseline c-peptide at 12 weeks and 48 weeks
Change of AGE(Advanced Glycation End Products) | Baseline, 12 weeks, 48 weeks
  Change from baseline AGE(Advanced Glycation End Products) at 12 weeks and 48 weeks
Change of CGM(Continuous Glucose Monitoring) | Baseline, 12 weeks, 48 weeks
  Change from baseline CGM(Continuous Glucose Monitoring) at 12 weeks and 48 weeks
Adverse events | 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hoyeon Chung, MD, PhD, Principal Investigator — Kyung Hee University Hospital at Gangdong
Locations (7):
- South Korea (7):
  - GangNeung Asan Hospital, Gangneung, Gangwondo
  - Inha University Hospital, Incheon
  - Kyung Hee University Hospital, Seoul
  - Soon Chun Hyang University Hospital Seoul, Seoul
  - Konkuk University Medical Center, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No